CLINICAL TRIAL: NCT06861517
Title: Deep Dictionaries for Feature Extraction in Context of Sparse Data for Electroencephalographic Signals from Brain-computer Interfaces
Brief Title: EEG-based Brain-computer Interface Database for Motor Rehabilitation
Status: Completed | Type: Observational
Sponsor: Jaime Alejandro Quiroga Forero (Other)
Responsible Party: Sponsor-Investigator, Jaime Alejandro Quiroga Forero, Principal Investigator, Universidad Nacional de Entre Rios
Organization: Universidad Nacional de Entre Rios (Other)
Other Study IDs: IS004678
Record Dates: First submitted 2025-02-24; First posted 2025-03-06 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-02

CONDITIONS: Healthy Adults
Keywords: EEG Signals Database; BCI; Effective Motor Activity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Healthly Volunteer

SUMMARY:
The human brain, as a processing center, controls bodily, cognitive, emotional and social functions, enabling perception, signal analysis and decision making. However, these functions can be affected by acquired brain injury (ABI), resulting from traumatic (blows to the head) or non-traumatic factors (tumors, strokes, infections, among others). Annually, about 55 million new cases of ABI are reported, with sequelae that can affect the quality of life of patients and their families. This scenario has driven research into tools to mitigate and recover lost capabilities. The Center for Rehabilitation Engineering and Neuromuscular and Sensory Research (CIRINS) of the Faculty of Engineering of the National University of Entre Ríos in Argentina has developed neuromuscular and sensory rehabilitation systems, with a focus on the innovation of motor rehabilitation tools using EEG-based brain-computer interfaces (BCI). These BCIs stand out for their economy and versatility, showing significant effects in the rehabilitation of motor functions. Challenges in BCI include signal complexity, artifacts, and inter-person variability, making it difficult to estimate user intent and extending calibration time. To mitigate these problems, strategies based on Deep Learning and dictionary learning have been proposed, which allow for sparse representations of data, being robust to noise and missing data, but with challenges in classification. The study proposes to develop a database of electroencephalographic signals applicable in the development of new algorithms for processing and feature extraction of this type of signals, contributing to the development of technology that supports rehabilitation processes.

ELIGIBILITY:
Inclusion Criteria:

* Willingness and ability to fully understand the purpose and scope of the experiment and to comply with the experiment instructions.
* Ability to easily distinguish visually the figures in the study.
* Ability to perform tasks that demand sustained concentration.

Exclusion Criteria:

* History of neurological diseases.
* Suffering from any type of musculoskeletal disorder that limits the motor skills necessary for the experiment.
* Having a significant hearing loss that prevents him/her from hearing the study instructions.
* Pregnancy.
* Lack of cooperation.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Volunteers of legal age and under 60 years of age, of any gender and without a history of neurological diseases
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2024-09-02 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Sensory motor rhythms power bands | Day 1
  The volunteer performs a movement task after a cue. A 32-channel EEG records signals following the 10-20 system and measures sensory-motor rhythm power bands.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Engineering, National University of Entre Ríos, Oro Verde, Entre Ríos Province, Argentina

IPD SHARING:
Plan to Share IPD: No
The study will focus on electroencephalography signals, therefore for now it is not considered relevant to include data from individual participants (IPD).

REFERENCES:
- See also: Publication about EEG Sensorimotor Rhythms — https://link.springer.com/chapter/10.1007/978-3-031-61973-1_1
- See also: Motor Intention in EEG-Based BCI — https://link.springer.com/chapter/10.1007/978-3-031-49407-9_10